CLINICAL TRIAL: NCT03545620
Title: Evaluation of Rescue Techniques After Failed Direct Laryngoscopy: A Multicentered Prospective Observational Study
Brief Title: Evaluation of Intubation Rescue Techniques on Management of Difficult Airway
Status: Completed | Type: Observational
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayse Zeynep Turan, Principle Investigator, Derince Training and Research Hospital
Other Study IDs: DerinceTRH-04
Record Dates: First submitted 2018-04-18; First posted 2018-06-04 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Difficult Intubation; Difficult Airway
Keywords: difficult airway; difficult intubation; videolaryngoscope; exchange catheter; fiberoptic bronchoscope; Laryngeal subglottic airway device; tracheostomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Difficult intubation,: Patients who underwent surgery under general anesthesia will be follow up. Patients predicted difficult intubation/airway or established difficult intubation/airway after anesthesia induction will be included. Which rescue technique will be used after unsuccessful direct laryngoscopy will be recorded.
  Interventions: Device: rescue technique

INTERVENTIONS:
Device: rescue technique — which rescue technique will be preferred while established/predicted difficult airway/intubation occurs in the operation room after failed direct laryngoscopy

SUMMARY:
When difficult airway/intubation occurs in the OR the anesthesiologist needs rescue techniques and equipment. The algorithms about management of the difficult airway don't provide adequate data. In current study researchers aim to determine most preferred rescue techniques and success rate of the chosen technique.

DETAILED DESCRIPTION:
In anesthesia setting Failed tracheal intubation, leading mortality and morbidity is very important. In operation room when a Difficult intubation occured with concurrent difficult mask ventilation rapid manipulation and quick decision are lifesaving. The Presence of assistant medical personnel or rescue equipment and crisis management of physician is crucial. In anesthesia practice when difficult airway occured rescue techniques are used to facilitate the intubation but difficult airway algorithms do not provide adequate information which rescue technique should be used in a state of emergency in OR thereby current trial was designed to determine which rescue techniques are used in everyday practice to manage difficult intubation, success and complication rates of chosen techniques.

Aim of the study

1. Most preferred rescue technique of the anesthesiologist When a difficult airway or difficult intubation ventilation occured
2. success rate of the chosen technique
3. Incidence of possible complications
4. Most preferred rescue technique of the anesthesiologist on presence of the difficult mask ventilation

ELIGIBILITY:
Inclusion Criteria:

* aged over 18 years
* patient underwent surgery under general anesthesia

Exclusion Criteria:

* pediatric patients
* patients who will intubate due to rapid serial intubation protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent surgery under general anesthesia over 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2017-12-03 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
which rescue technique will be chosen by the anesthesiologist after failed direct laryngoscopy | Participants will be followed for the duration of anesthesia and after induction, an expected average of 1 hour
  In case of a difficult airway situation after anesthesia induction patients will be enrolled to the study. Researchers will observe the case and record the chosen rescue technique such as video laryngoscope, supraglottic airway device, fiberoptic intubation or tracheostomy. Here the researchers aim to observe the preferred rescue method of providing an intact airway.

SECONDARY OUTCOMES:
the success rate of chosen technique for providing an intact airway | Participants will be followed for the duration of anesthesia and after induction, an expected average of 1 hour
  Tracheal intubation or supraglottic airway device insertion period will be observed. When end tidal CO2 will be seen on the monitor patient's airway will be accepted as successfully provided. .
Complications due to intubation | Participants will be followed for the duration of anesthesia and after induction, an expected average of 12 hour
  intubation period will be observed and patients will be followed up for complications including throat pain, trauma (pharyngeal, laryngeal, teeth, palate) hypoxemia, death,
Determination of the most preferred rescue technique for the anesthesiologists during difficult airway management. | Participants will be followed for the duration of anesthesia and after induction, an expected average of 1 hour
  The researchers aim to determine the most preferred rescue technique for the anesthesiologists during difficult airway management.Researchers will observe the case and record the chosen rescue technique such as video laryngoscope, supraglottic airway device, fiberoptic intubation or tracheostomy. Here the researchers aim to observe the preferred rescue method of providing an intact airway.

CONTACTS AND LOCATIONS:
Overall Officials: mehmet yilmaz, Study Director — Sağlık Bilimleri Üniversitesi Kocaeli Derince Eğitim ve Araştırma Hastanesi
Locations (4):
- Turkey (Türkiye) (4):
  - Haydarpasa Numune Researh and Training Hospital, Istanbul
  - Marmara University School of Medicine, Istanbul
  - Derince Research and Training Hospital, Kocaeli
  - Kocaeli University School of Medicine, Kocaeli